CLINICAL TRIAL: NCT03663660
Title: Design of an Organizational Infrastructure Pediatric Plan to Deal With Bronchiolitis Epidemics: Impact on Length of Stay and Quality of Care in a Tertiary Care Regional Hospital
Brief Title: Organizational Infrastructure Pediatric Plan in Bronchiolitis Epidemics
Acronym: OIPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0174
Record Dates: First submitted 2018-06-20; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-06

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Health care; Organizational change; children; Epidemic; cost
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before the OIPP: Period 1 : Children hospitalized before the OIPP implementation
- after the OIPP implementation: Period 2 :Children hospitalized after the OIPP implementation
  Interventions: Other: Organizational infrastructure pediatric plan (OIPP)

INTERVENTIONS:
Other: Organizational infrastructure pediatric plan (OIPP) — Restructuration of the hospital sectors with a stratification of health care into 4 levels.
  Groups: after the OIPP implementation

SUMMARY:
Acute bronchiolitis is a frequent respiratory viral infection of infants, responsible for 460,000 new cases per year in France. Over the years, the number of hospitalizations during the epidemic season appears to be increasing. Bronchiolitis epidemics lead to recurrent hospital disruption. The current trend towards a reduction of hospital beds is exacerbating the pressure on bronchiolitis epidemics on healthcare systems.

In this context, the pediatric departments of Montpellier University Hospital, France, designed in 2014 a common organizational infrastructure pediatric plan (OIPP) to to adapt to these multiple constraints while respecting the quality of care.

This plan includes a referral flowchart for hospitalized children, an increase in medical and paramedical staff and a restructuring of the pediatric units, with a specific stratification into 4 levels of care.

The study aims to assess the impact of our OIPP on the overall length of stay for children hospitalized for bronchiolitis. The investigator also intend to measure the impact of the OIPP on the length of stay within each unit, the number of transfers from one unit to the other and the number of readmissions within 30 days after hospital discharge. The cost of the implementation of the OIPP in the structure will be analyzed.

DETAILED DESCRIPTION:
The investigator compared data between two periods of time, e.g. the two consecutive years before the beginning of the OIPP (winters 2012-2013 and 2013-2014) and two first years after the beginning of the OIPP (winters 2015-2016 and 2016-2017).

ELIGIBILITY:
Inclusion criteria:

* age < 2 years
* hospitalization for bronchiolitis

Exclusion criteria:

* None

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Chidren under 2 years hospitalized for bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 1636 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Overall hospital length of stay | 1 year
  Overall hospital length of stay

SECONDARY OUTCOMES:
Hospitalization rate in ICU | 1 year
  Rate of hospitalization in intensive care unit
Readmissions within 30 days after hospital discharge | 30 days
  Number of readmissions in our hospital in the 30 days after hospital discharge
Transfer rate between units | 1 year
  Transfer rate between units
Cost of the OIPP implementation in our institution | 1 year
  Cost of the OIPP implementation in our institution

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Lavilledieu D, Abassi H, Mercier G, Guiraud M, Chaffaut GD, Milesi C, Cambonie G, Gavotto A, Jeziorski E, Amedro P. Implementation of an organizational infrastructure paediatric plan adapted to bronchiolitis epidemics. J Infect Public Health. 2020 Feb;13(2):167-172. doi: 10.1016/j.jiph.2019.07.007. Epub 2019 Aug 2. PMID 31378693